CLINICAL TRIAL: NCT06744699
Title: A Retrospective Observational Medical Dossier-based Study to Assess Gastrointestinal Discomfort and Infections in Healthy Term Infants
Brief Title: Assessment of Gastrointestinal Discomfort and Infections in Healthy Term Infants
Acronym: MESK-1
Status: Active, not recruiting | Type: Observational
Sponsor: Ausnutria Hyproca B.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: P24-151
Record Dates: First submitted 2024-11-19; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Gastrointestinal Symptoms; Infection; Allergy Symptoms; Growth
Keywords: infant; retrospective; medical dossier-based study; GI symptoms; infection symptoms; allergy symptoms; type of feeding; growth
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Formula-fed infants: Formula-fed infants either goat milk-based infant formula or cow's milk-based infant formula
  Interventions: Other: Infants fed goat milk-based infant formula

INTERVENTIONS:
Other: Infants fed goat milk-based infant formula — Type of infant feeding during the age of 0-12 months
  Other Names: Infants fed cow's milk based infant formula; Infants breastfed / human milk feeding

SUMMARY:
A retrospective observational medical dossier-based study to assess gastrointestinal discomfort and infections in healthy term infants

DETAILED DESCRIPTION:
Gastrointestinal (GI) symptoms like regurgitation, unexplained crying and stool issues (diarrhoea or constipation) are common in young infants <4 months of age due to an immature gut epithelial barrier, immune system and microbiota, with studies indicating prevalences ranging from 25.9%-78%. This retrospective observational medical dossier-based study is designed to determine the occurrence of GI symptoms in healthy term formula-fed infants to confirm reported prevalence of mild GI symptoms by HCPs in Middle East (74%). As a secondary objective, the improvement of confirmed GI symptoms when switched before 4 months of age from a CMF to GMF will be determined. Based on the results of a previous study in infants with confirmed GI symptoms, it is expected that fewer GI symptoms will be scored in medical dossiers of infants after switching from CMF to GMF, with HM as a reference group. Other secondary objectives of this study are to explore differences between healthy term infants that were fed GMF compared to infants fed CMF or HM on immune related outcomes such as infections and allergies, medication use related to infections and/or gastrointestinal discomfort and/or allergies, number of clinic visits, adequate growth and reason of changing infant formula.

ELIGIBILITY:
Inclusion Criteria:

* Either exclusively formula fed (GMF or CMF; consumption of HM ≤2 weeks is allowed for formula fed infants) OR exclusively breastfed before introduction of complementary feeding.
* Age 12-24 months of age to ensure collection of recent data.
* If required by local regulation or guidelines, written informed consent (ICF) from Investigator (or parent(s) and/or caregiver(s)* aged ≥18 years).
* Singleton, term infants (gestational age ≥ 37 weeks and ≤ 42 weeks).
* At least 6 reported visits to the doctor between 0-12 months of age.

Exclusion Criteria:

* Consumed hydrolysed infant formula or other specialty formulas.
* Any current or previous illnesses/conditions and/or known congenital diseases or malformations which could interfere with the study outcomes, as per Investigator's clinical judgement.
* Participation in any clinical trial during first year of life.
* For formula-fed infant, no switch in feeding type after 4 months of age is allowed.

Max Age: 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population consists of 300 healthy term infants with medical dossiers covering the period of 0-12 months of age and at least 6 clinic visits.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
To investigate the occurrence of symptoms related to GI discomfort in formula-fed infants in the Gulf region | retrospective infants from 0 - 12 months of age
  To determine the number of symptoms related to GI discomfort in formula-fed infants between 0-12 months of age

CONTACTS AND LOCATIONS:
Locations (3):
- Saudi Arabia (3):
  - Al Emies hospital, Jizan
  - Mana GH Jubail, Jubail
  - AlAhmady Hospital, Madinah

IPD SHARING:
Plan to Share IPD: No